CLINICAL TRIAL: NCT06158074
Title: Efficacy of Electrical Pudendal Nerve Stimulation and Sacral Neuromodulation in Treating Non-obstructive Neurogenic Urinary Retention: A Nonrandomized Clinical Trial
Brief Title: Efficacy of Electrical Pudendal Nerve Stimulation and Sacral in Treating Non-obstructive Neurogenic Urinary Retention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Institute of Acupuncture, Moxibustion and Meridian (Other)
Collaborators: Shanghai Pudong Hospital of TCM (Unknown); Shanghai Yueyang Integrated Medicine Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-099
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2023-12

CONDITIONS: Urinary Retention
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EPNS group (Experimental)
  Interventions: Procedure: electrical pudendal nerve stimulation
- SNM group (Active Comparator)
  Interventions: Procedure: sacral neuromodulation

INTERVENTIONS:
Procedure: electrical pudendal nerve stimulation — The patient was positioned prone post-micturition. Long needles (0.40 Х 100 mm) were inserted perpendicularly, 1 cm bilateral to the sacrococcygeal joint, to a depth of 80-90 mm, eliciting sensations referred to the urethra or anus. The lower points, 1 cm bilateral to the coccyx tip, received oblique insertion of longer needles (0.40 Х 125 mm) toward the ischiorectal fossa (90-110 mm depth), inducing sensations precisely to the urethra. Connected to a G6805-2 Multi-Purpose Health Device, the ipsilateral needles created an electric loop, with the upper as anode and lower as cathode. Direct electrical stimulation (2.5 Hz, 25~35 mA) for 60 minutes targeted the pudendal nerve, thrice weekly for a total of 4 weeks.
  Arms: EPNS group
Procedure: sacral neuromodulation — In the prone position, patients undergo sacral nerve root localization through MRI and CT fusion analysis. A 3D-printed sacral foramen puncture template is crafted for precision. Using local anesthesia, a 20G needle at a 60° angle enters the S3 sacral foramen along the template. A temporary stimulator, delivering square waves (14-35 Hz, 210-360 μs), tests motor and sensory responses to confirm accuracy. Self-fixating electrodes are then implanted, validated, and tunneled subcutaneously. External connection to a temporary stimulator provides a 4-week therapeutic experiential stimulation.Patients are administrated by antibiotics peri-operatively to prevent lead site infection.
  Arms: SNM group

SUMMARY:
To observe the clinical effects and make a comparative study between efficacy of electrical pudendal nerve stimulation (EPNS) and sacral neuromodulation (SNM) , evaluate the advantages of EPNS in the treatment of neurogenic non-obstructive urinary retention, and provide a new method for the treatment of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Non-mechanical obstructive urinary retention occurs following relevant neurological system disorders (spinal cord injury, spina bifida，myelitis, cervical/thoracic disk disease, lesion following spinal anesthesia/spine surgery,lumbar/sacral spine intervertebral disc diseases, spinal stenosis, iatrogenic pelvic nerve lesions, sacral agenesis, peripheral neuropathy due to diabetes mellitus).
* With normal upper urinary tract function.
* Other therapies and medications potentially affecting the assessment of this therapy have been discontinued for at least two weeks before the interventional procedure.
* Patient with good compliance who is capable of cooperating with the follow-up requirements

Exclusion Criteria:

* Patients with any suprapontine and pontine lesions
* Pregnant or lactating women
* Individuals whose symptoms show significant improvement after pharmaceutical and adjunctive therapy
* Individuals with concurrent acute or chronic prostatitis, prostate cancer, or conditions such as bladder neck stenosis, urethral stricture, or urethral injury
* High pathological risk factors (e.g., lymph node metastasis, resection margin involvement, bulky tumors)
* Individuals with concomitant obstructive urinary retention

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Percent change in pre-post treatment post-voiding residual urine volume (PVR ) | baseline (T0), mid-treatment (T1; after 6 EPNS sessions or 2 weeks of SNM), and (T2; after 12 EPNS sessions or 4 weeks of SNM)
  Bladder PVR is measured by ultrasound.Percent change in pre-post treatment PVR is calculated as (baseline PVR - post-treatment PVR) / baseline PVR × 100%.

SECONDARY OUTCOMES:
Absolute post-voiding residual volume (PVR) at the end of treatment; International Consultation on Incontinence Questionnaire-Lower Urinary Tract Symptoms (ICIQ-LUTS) and the quality of life (ICIQ-LUTSqol) score. | Mid-treatment (T1; after 6 EPNS sessions or 2 weeks of SNM), and (T2; after 12 EPNS sessions or 4 weeks of SNM)
  Absolute PVR <50 mL is regarded as a clinically meaningful target; ICIQ-LUTS and ICIQ-LUTSqol are two patient-reported outcomes

OTHER OUTCOMES:
achievement of ≥50% PVR improvement rate and composite achievement (requiring both PVR <50 mL and ≥50% PVR improvement rate) | mid-treatment (T1; after 6 EPNS sessions or 2 weeks of SNM), and (T2; after 12 EPNS sessions or 4 weeks of SNM)
  Binary clinical targets (achievement / failure)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai research institute of acupuncture and meridian, Shanghai, China

IPD SHARING:
Plan to Share IPD: No